CLINICAL TRIAL: NCT00582790
Title: Phase II Study of Interleukin-2 in Combination With Zoledronic Acid in Patients With Untreated Metastatic Renal Cell Carcinoma
Brief Title: Study of IL2 in Combination With Zoledronic Acid in Patients With Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC 2003-170; CO03805; A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2013-03

CONDITIONS: Kidney Cancer
Keywords: Renal Cell Cancer; Metastatic
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Interleukin-2; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Interleukin-2 subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles in combination with Zoledronic acid IV on day 1 of every 4 week (28 days) cycle.
  Interventions: Drug: IL2; Drug: Zoledronic acid

INTERVENTIONS:
Drug: IL2 — Interleukin-2 will be given at a starting dose of 7 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles.
  Other Names: Interleukin-2
Drug: Zoledronic acid — Zoledronic acid will be given on day 1 intravenously over 15 or 30 minutes starting at 400mcg. If no significant increase in gamma delta-T cell augmentation is seen, the dose of zoledronic acid will be increased in the subsequent cycle up to a maximum dose of 3mg.
  Other Names: Zometa

SUMMARY:
This study is being done to see if we can improve the response of Interleukin-2 by adding Zoledronic acid. The effectiveness of the combination of drugs in kidney cancer is unknown and will be investigated in this study. In particular, this study will evaluate the effect of this combination on kidney cancer and will also examine the safety and side effects of IL-2 with Zoledronic acid.

DETAILED DESCRIPTION:
The purpose of this research is to evaluate the antitumor response of low-dose Interleukin-2 in combination with Zoledronic acid on subjects with previously untreated, unresectable metastatic renal cell carcinoma. Also, the study will assess the tolerability, safety, pharmacodynamic effects, and immunologic effects of low-dose Interleukin-2 in combination with Zoledronic acid on angiogenesis inhibition and anti-metastatic potential by measuring serum/plasma angiogenic/metastatic factor levels and by quantitating changes in cytokine expression, antigen-specific T-cell immune responses, and peripheral gd T-cell frequency and function.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma with metastasis.
* Must have measurable disease.
* No prior cytokine, chemotherapy, hormonal, or other immuno-based therapies (including vaccine or cellular based) for their renal cancer is allowed. No prior use of bisphosphonates will be allowed. One prior experimental therapy will be permitted as long as > 4 weeks have passed since last drug administration.
* ECOG performance status 0 or 1
* Adequate cardiac function by history.
* Pulse-oximetry > 92% on room air.

Exclusion Criteria:

* Radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Known brain metastases
* Any history of an autoimmune disease (ie. psoriasis, inflammatory bowel disease, etc) must receive clearance by the investigator before being permitted on study due to the potential worsening of those disorders from IL-
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* History of myocardial infarction or hospitalization for congestive heart failure within 12 months of enrollment.
* History of prior malignancy (except basal cell carcinoma resected with curative intent) unless resected or treated with curative intent and disease free for > 5 years.
* Any history of seizures given increased seizure risk with IL-2.
* Organ allograft (transplant) recipients will be excluded given absolute contraindication with IL-2 therapy.
* Pregnant women are excluded
* Patients on systemic steroids (oral or IV) will not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2003-08; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to accrual on 09/30/2003 and closed to accrual on 08/05/2008. Recruitment occured in a medical clinic.
Groups:
- Zoledronic Acid and Interleukin-2: Patients 1-6: Zometa at 4mg intravenously on day 1 of each 28-day cycle and IL-2 at a starting dose of 7 MU/m2/day by subcutaneous injection days 1-5, weekly in weeks 1 through 3 of each cycle.
  patients 7, 8 and 9: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles.
  The last patients: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles and dose escalation of zometa.
Period: Overall Study
Arm/Group | Zoledronic Acid and Interleukin-2
Started | 12 (only 11 of the 12 patients received study treatment.)
Completed | 11
Not Completed | 1
Not completed — Rapid progression of disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid and Interleukin-2
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antitumor Response With Low-dose Interleukin-2 in Combination With Zoledronic Acid
Description: Anti-tumor response was measured per RECIST criteria (V1.0) and assessed by chest/abdomen/pelvis CT: Complete Response (CR), disappearance of all target lessions; Partial Response (PR), >=30% decrease in the sum of the longest diameter (LD) of target lesions; Stable Response (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started.
Time Frame: CT scans obtained at baseline, then every 2 cycles
Population: Anti tumor response was measured in those patients who completed at least 1 cycle of study treatment 4 subjects did not complete 1 cycle of treatment.
Measure: Number; unit: participants
Groups:
- IL2 and Zoledronic Acid: Patients 1-6: Zometa at 4mg intravenously on day 1 of each 28-day cycle and IL-2 at a starting dose of 7 MU/m2/day by subcutaneous injection days 1-5, weekly in weeks 1 through 3 of each cycle.
  patients 7, 8 and 9: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles.
  The last patients: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles and dose escalation of zometa.
Arm/Group | IL2 and Zoledronic Acid
Number analyzed (Participants) | 8
participants | 5

2. Secondary Outcome: Number of Participants With Overall Survival and Progression-free Survival at 24 Weeks
Description: All 12 patients were followed for survival until death. 8 participants who received more than one cycle of treatment and who were considered evaluable for response were followed until time to progression. Disease progression was determined by CT scans of the chest/abdomen/pelvis obtained every 2 cycles and based on RECIST version 1.0. Progression is defined using RECIST (V1.0) at least a 20% increase in the sum of the longest diameter (LD)of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: Time frame is from study entry until time to disease progression and time to death, up to 50 months
Population: 8 of the 12 participants who received more than 1 cycle of therapy and were considered evaluable for time to progression. All 12 were evaluated for survival
Measure: Number; unit: participants
Arm/Group | IL2 and Zoledronic Acid
Number analyzed (Participants) | 12
participants | 5 [4 to 33]

3. Secondary Outcome: Number of Participants With Toxicities
Description: Patients were observed for toxicities. The National Cancer Institute Common Terminology Criteria Version 2.0 was used to categorize and report adverse events.
Time Frame: Baseline to 30 days after last dose of study treatment
Population: Patients who received at least one dose of study medication. One of the 12 patients never received study medication so only 11 were evaluable for toxicity
Measure: Number; unit: participants
Arm/Group | IL2 and Zoledronic Acid
Number analyzed (Participants) | 11
participants | 11

4. Secondary Outcome: Number of Participants With Immunologic Responses
Description: Blood was collected to analyze T-cell populations from all patients prior to treatment on day 1 of cycles 1 and 2, and days 4 and 8 of cycles 1 and 2. Changes in gamma delta T-cell population and CD3 T-cell populations were reported.
Time Frame: baseline to cycle 2 day 8
Population: One patient did not receive study treatment and so was not included in the analysis.
Measure: Number; unit: participants
Groups:
- Low-dose IL2 and Zoledronic Acid: Patients 1-6: Zometa at 4mg intravenously on day 1 of each 28-day cycle and IL-2 at a starting dose of 7 MU/m2/day by subcutaneous injection days 1-5, weekly in weeks 1 through 3 of each cycle.
  patients 7, 8 and 9: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles.
  The last patients: IL-2 at a dose of 1 MU/m2/day by subcutaneous injection days 1-5, on weeks 1 through 3, in four week (28 days) cycles and dose escalation of zometa.
Arm/Group | Low-dose IL2 and Zoledronic Acid
Number analyzed (Participants) | 11
participants | 0

ADVERSE EVENTS:
Time Frame: Study period: 2003 to 2006. Adverse events were collected from time of study treatment to 30 days post treatment.
Description: Adverse events listed are those with at least possibly related. All SAE's are reported regardless of whether or not they were felt related to study procedures.
Arm/Group | Zoledronic Acid and Interleukin-2
Serious Adverse Events (participants affected / at risk) | 2/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid and Interleukin-2 (N=11)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Creatinine (Renal and urinary disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid and Interleukin-2 (N=11)
Hypotension (Cardiac disorders) | 4 (5)
Creatinine (Renal and urinary disorders) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomitting (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Myalgias (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgias (Musculoskeletal and connective tissue disorders) | 4 (5)
Bone pains (Musculoskeletal and connective tissue disorders) | 5 (5)
Hand edema (Musculoskeletal and connective tissue disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Infection NOS (Infections and infestations) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
SGPT (ALT) (Hepatobiliary disorders) | 4 (4)
SGOT (AST) (Hepatobiliary disorders) | 4 (4)
GGT (Hepatobiliary disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3)
Headache (Nervous system disorders) | 4 (4)
Anxiety/Depression (Psychiatric disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry Eye (Eye disorders) | 1 (2)
Weight Loss (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Fatigue (General disorders) | 6 (9)
Chills (General disorders) | 9 (9)
Fever (General disorders) | 7 (7)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Non-Cardiac Chest (General disorders) | 1 (4)
Myalgias/Arthralgias (General disorders) | 5 (8)
Musculocskeletal (General disorders) | 7 (7)
injection site reaction (General disorders) | 7 (7)
Taste changes (General disorders) | 2 (2)
Thyroiditis (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No